CLINICAL TRIAL: NCT06108713
Title: The Effect of Juggling Training on Some Cognitive Functions and Coordination Abilities in Older People.
Brief Title: The Influence of Juggling on Selected Cognitive Functions and Postural Stability Variables.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 106/21
Record Dates: First submitted 2023-10-13; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Aging; Cognitive Change
Keywords: cognitive functions; postural stability; proprioception; elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Addition of juggling (Experimental): Group taking part in juggling exercise protocol in a crossover regimen.
  Interventions: Other: Addition of juggling
- Without addition of juggling (No Intervention): Group not taking part in juggling exercise protocol in a crossover regimen.

INTERVENTIONS:
Other: Addition of juggling — Participants will not change ther daily activities, and participate in juggling intervention lasted 4 weeks and consisted of 12 meetings (3 trainings per week), each lasting 45 minutes.
  Arms: Addition of juggling

SUMMARY:
The purpose of the study is to verify the effect of juggling exercises on selected cognitive functions (reaction time, attention) and postural stability variabilities (based on center of pressure signal) in two different protocols: [1] a randomised crossover study design, [2] a randomised repeated measurement design.

DETAILED DESCRIPTION:
Juggling is a form of exercise, that can engage humans, both cognitively and physically. One of the positive aspects of taking up this form of exercise is the growing evidence indicating that juggling improves the well-being of exercisers. Most importantly, the juggling intervention causes an increase in the volume of the gray matter and white matter in the human brain, and thus shows potential for neuroplasticity. In addition, unhealthy aging is observed nowadays, which causes both physical and cognitive decline in daily functioning, further interfering with the elderly's ability to perform daily activities. Therefore, the addition of juggling exercises may have a positive effect on the changes that occur with aging.

However, currently there are hardly any data on the juggling effect on cognitive functions and on postural stability. Therefore, the study aims to examine the effect of juggling exercises on selected cognitive functions and postural stability variables in two different randomised trials.

ELIGIBILITY:
Inclusion Criteria:

* physically active
* over 65 years old
* with no injuries of pathologies involving the upper limb
* without neurological issues
* with no significant visual impairments

Exclusion Criteria:

* mixed or left-handedness
* sedentary lifestyle
* prior experience in juggling
* under or above the required age
* contraindications to physical activity

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Velocity of center of pressure assessed with AMTI force plate | Assessment of the velocity of center of pressure will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Postural stability variable based on center of pressure signal. Velocity of center of pressure will be presented in centimeters per seconds.
Area 95 percentile assessed with AMTI force plate | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Postural stability variable based on center of pressure signal. Area 95 percentile will be presented in square centimetres.
Medio-lateral range of sway assessed with AMTI force plate | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Postural stability variable based on center of pressure signal. Medio-lateral range of sway will be presented in centimeters.
Anterior-posterior range of sway assessed with AMTI force plate | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Postural stability variable based on center of pressure signal. Anterior-posterior range of sway will be presented in centimeters.
Effective value of medio-lateral velocity assessed with AMTI force plate | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Postural stability variable based on center of pressure signal. Effective value of medio-lateral velocity of sway will be presented in centimeters per seconds.
Effective value of anterior-posterior velocity assessed with AMTI force plate | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Postural stability variable based on center of pressure signal. Effective value of anterior-posterior velocity of sway will be presented in centimeters per seconds.
Absolute error of elbow joint position accuracy assessed with electrogoniometers | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Proprioception ability. Measured in degrees of flexion.
Variable error of elbow joint position accuracy assessed with electrogoniometers | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Proprioception ability. Measured in degrees of flexion.
Constant error of elbow joint position accuracy assessed with electrogoniometers | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Proprioception ability. Measured in degrees of flexion.
Root mean square error of elbow joint position accuracy assessed with electrogoniometers | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Proprioception ability. Measured in degrees of flexion.

SECONDARY OUTCOMES:
Simple reaction time assessed with reaction time test in Vienna Test System | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Selected cognitive function - simple reaction time (one visual stimulus, reaction to one visual stimulus) measured in milliseconds.
Complex reaction time assessed with reaction time test in Vienna Test System | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Selected cognitive function - choice reaction time (two visual stimuli, reaction to one visual stimulus) measured in milliseconds.
Decision time assessed with reaction time test in Vienna Test System | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Selected cognitive function - decision time (difference between complex reaction time and simple reaction time variables) measured in milliseconds.
Motor time assessed with reaction time test in Vienna Test System | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Selected cognitive function - motor reaction time (time of movement during both simple and complex reaction time tests) measured in milliseconds.
Time of correct rejections assessed with cognitrone test in Vienna Test System | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Selected cognitive function - one variable of attention measured in seconds.
Time of correct acceptance assessed with cognitrone test in Vienna Test System | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Selected cognitive function - one variable of attention measured in seconds.
Number of correct acceptance assessed with cognitrone test in Vienna Test System | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Selected cognitive function - one variable of attention measured in unity values.
Duration of test assessed with cognitrone test in Vienna Test System | Assessment will be carried out up to three days before juggling/no juggling periods, and also up to three days after juggling/no juggling periods. Measurements will be taken at a total of four time points.
  Selected cognitive function - one variable of attention measured in seconds.
Physical activity level assessed with a CHAMPS questionnaire | Assessment will be carried out up to three days after juggling/no juggling periods. Measurements will be taken at a total of two time points.
  Assesment of physical activity level with a CHAMPS questionnaire. Results presented as frequency of total physical activity and caloric expenditure per week.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Malik, MSc, Principal Investigator — Department of Physical Activity and Health Promotion Science
Locations (1):
- Poznan University of Physical Education, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malik J, Glowka N, Jelonek W, Maciaszek J. The effect of juggling on the proprioceptive and attentional abilities among older women. Front Public Health. 2024 Oct 2;12:1386981. doi: 10.3389/fpubh.2024.1386981. eCollection 2024. PMID 39416927
- [Derived] Malik J, Glowka N, Jelonek W, Stemplewski R, Maciaszek J. Effect of a juggling-based physical activity on postural stability, reaction time, and attention focus in older adults: a randomized crossover study. Eur Rev Aging Phys Act. 2024 May 31;21(1):15. doi: 10.1186/s11556-024-00351-w. PMID 38822245